CLINICAL TRIAL: NCT07307144
Title: Fractalkine and CX3CR1 Dynamics in Gingivitis and Periodontitis Before and After Therapy
Brief Title: Fractalkine-CX3CR1 Axis in Periodontal Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Giresun University (Other)
Responsible Party: Principal Investigator, Zeynep Pınar Yucel, Assoc. Prof., Giresun University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: OMU KAEK 2022/85; SAĞ-BAP-A-240222-47 (Other Grant/Funding Number: Giresun University Scientific Research Projects Coordination Unit)
Record Dates: First submitted 2025-12-13; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Periodontitis; Gingivitis; Inflammation Biomarkers
Keywords: periodontitis; gingivitis; gingival crevicular fluid
MeSH Terms: conditions — Periodontitis; Gingivitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- stage 3 periodontitis (Active Comparator): GCF samples were collected at baseline and at 1 and 3 months after treatment from periodontitis patients.
  Interventions: Other: Non-surgical periodontal treatment
- Gingivitis (Active Comparator): GCF samples were collected at baseline and at 1 and 3 months after treatment from gingivitis patients.
  Interventions: Other: Non-surgical periodontal treatment
- Periodontally healthy controls (No Intervention): GCF samples were collected from periodontally healthy controls at baseline for once.

INTERVENTIONS:
Other: Non-surgical periodontal treatment — Scaling and root planing, oral hygiene education and motivation.
  Arms: Gingivitis; stage 3 periodontitis

SUMMARY:
This study aimed to evaluate gingival crevicular fluid (GCF) levels of fractalkine/CX3CL1 and CX3CR1 in patients with gingivitis and periodontitis before and after non-surgical periodontal therapy.

DETAILED DESCRIPTION:
Thirty stage 3 periodontitis, thirty gingivitis and thirty periodontally healthy individuals were enrolled in the study. Clinical periodontal measurements were recorded; gingivitis and periodontitis patients underwent non-surgical periodontal treatment, and GCF samples were collected at baseline and at 1 and 3 months after treatment. CX3CL1 and CX3CR1 were determined by ELISA.

ELIGIBILITY:
Inclusion Criteria:

1. 25-50 years of age
2. having at least 20 natural teeth, excluding third molars
3. having no systemic disease
4. non-smokers
5. criteria for healthy control group: BOP < 10% and PD ≤ 3 mm without clinical attachment loss or radiographic sign of alveolar bone destruction
6. criteria for stage 3 periodontitis group: interdental CAL ≥ 5 mm at least 2 non-adjacent teeth, PD ≥ 6 mm and radiographic bone loss extending to the mid-third of the root or beyond.

Exclusion Criteria:

1. having any systemic diseases,
2. smoking
3. current pregnancy or lactation
4. a history of periodontal treatment in the past 6 months
5. using antibiotic, anti-inflammatory drugs or any other drugs within the past 6 months.

Ages: 25 Years to 47 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2022-05-15 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2023-12-10 (Actual)

PRIMARY OUTCOMES:
Changes in the levels of biochemical parameters | Baseline and 1 and 3 months after treatment
  The levels of Fractalkine and CX3CR1 before and after periodontal treatment in gingivitis and periodontitis patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Giresun University, Giresun, Turkey, Turkey (Türkiye)